CLINICAL TRIAL: NCT02491008
Title: Novel Biomarkers and Skeletal Outcomes Associated With Subclinical Thyroid Dysfunction: a Prospective Evaluation and Impact of Treatment
Brief Title: Novel Biomarkers and Skeletal Outcomes Associated With Subclinical Thyroid Dysfunction
Acronym: TRUST BONE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 162/11_3; SNF 320030_150025 (Other Grant/Funding Number: SNF)
Record Dates: First submitted 2015-07-02; First posted 2015-07-07 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Thyroid Dysfunction; Bone Mineral Density; Osteoporosis; Fractures, Bone
Keywords: Thyroid Dysfunction; Bone mineral density; Osteoporosis; Fractures, Bone; Randomized Controlled Trial
MeSH Terms: conditions — Osteoporosis; Fractures, Bone | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug: Levothyroxine (Experimental): The intervention will start with Levothyroxine 50 mcg daily (reduced to 25 mcg in subjects <50 kg of body weight or if known coronary heart disease - previous myocardial infarction or symptoms of angina pectoris) vs. matching placebo; at 3 months, if the serum TSH level is <0.4 mU/L, dose will be reduced by 25 mcg; TSH >=0.4 and <4.6 mU/L, no change to dose; TSH >=4.6 mU/L, additional 25 mcg. The process will be repeated at 12 months, then annually; mock titration will be performed in the placebo group. The maximum possible dose of Levothyroxine which will be prescribed is 150 mcg (after 4 increments of 25 mcg at 3 months, 1, 2, 3 years; from the starting dose of 50 mcg).
  Interventions: Drug: Levothyroxine
- Drug: Placebo (Placebo Comparator): Control patients will obtain a placebo pill of the same characteristics as the intervention drug, and mock titration will be carried out identically to the intervention drug.
  Pharmaceutical composition of placebo (100 mg): Lactose monohydrate 66 mg, Maize starch 25 mg, Gelatin 5 mg, Croscarmellose sodium 3.5 mg, Magnesium stearate (vegetable source) 0.5 mg.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levothyroxine — The intervention will start with Levothyroxine 50 mcg daily (reduced to 25 mcg in subjects <50 kg of body weight or if known coronary heart disease - previous myocardial infarction or symptoms of angina pectoris) vs. matching placebo; at 3 months, if the serum TSH level is <0.4 mU/L, dose will be reduced by 25 mcg; TSH >=0.4 and <4.6 mU/L, no change to dose; TSH >=4.6 mU/L, additional 25 mcg. The process will be repeated at 12 months, then annually; mock titration will be performed in the placebo group. The maximum possible dose of Levothyroxine which will be prescribed is 150 mcg (after 4 increments of 25 mcg at 3 months, 1, 2, 3 years; from the starting dose of 50 mcg).
  Arms: Drug: Levothyroxine
Drug: Placebo — Control patients will obtain a placebo pill of the same characteristics as the intervention drug, and mock titration will be carried out identically to the intervention drug.
  Pharmaceutical composition of placebo (100 mg): Lactose monohydrate 66 mg, Maize starch 25 mg, Gelatin 5 mg, Croscarmellose sodium 3.5 mg, Magnesium stearate (vegetable source) 0.5 mg.
  Arms: Drug: Placebo

SUMMARY:
Thyroid hormone is a key regulatory hormone for a range of physiological systems, including the skeleton. Previous studies have suggested that subclinical thyroid dysfunction (SCTD) may be associated with deleterious skeletal effects. However, controversy persists on the clinical relevance of SCTD as well as on optimal thresholds for treatment. Available data have substantial limitations: 1) limited prospective data are available to assess the associations between SCTD and non-cardiovascular outcomes, such as fractures 2) lack of data from large RCTs to investigate the pathophysiological mechanisms of associations between thyroid hormone and bone loss. The aim of the study is to examine the relationship between subclinical hypothyroidism and thyroid hormone replacement in regard to skeletal fragility, bone mineral density (BMD), bone loss and metabolism, and the risk of fractures in elderly participants. The listed parameters will be assessed by dual energy X ray absorptiometry (DXA) and novel bone imaging techniques at baseline, at 1 year of follow-up. The study will be nested in the TRUST trial (clinicaltrials.gov ID: NCT01660126), and will make use of its study infrastructure to determine bone biomarkers from biospecimens at baseline, and at 1 year of follow-up from 145 Swiss participants with persistent subclinical hypothyroidism randomized to either thyroxine or placebo in Bern and Lausanne.

DETAILED DESCRIPTION:
Background

Thyroid hormone is a key regulatory hormone for other physiological systems, including the skeleton. Previous studies have suggested that SCTD may be associated with deleterious skeletal effects. However, controversy persists on the clinical relevance of SCTD as well as on optimal thresholds for treatment. Available data have substantial limitations: 1) limited prospective data are available to assess the associations between SCTD and non-cardiovascular outcomes, such as fractures 2) lack of data from large RCTs to investigate the pathophysiological mechanisms of associations.

Objective

To examine, within a large RCT of elderly participants with subclinical hypothyroidism (the TRUST trial), the impact of thyroxine therapy on the association between SCTD and skeletal fragility, bone mineral density (BMD), bone loss and metabolism, and the risk of fractures.

Methods

The existing trial infrastructure (TRUST thyroid trial-Euresearch FP7,clinicaltrials.gov ID: NCT01660126) will be utilized to collect biospecimens from the 145 Swiss participants with persistent subclinical hypothyroidism randomized to either thyroxine or placebo in Bern and in Lausanne. The assessment is performed by means of dual energy X ray absorptiometry (DXA) and peripheral quantitative computed tomography (pqCT) as a novel bone imaging technique at baseline, and at 1 year of follow-up. In parallel, bone turnover markers in the blood plasma will be measured at baseline and at 1 year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling patients aged >= 65 years with subclinical hypothyroidism
* Written informed consent

Exclusion Criteria

* Subjects currently under levothyroxine or antithyroid drugs (amiodarone, lithium)
* Recent thyroid surgery or radio-iodine (within 12 months)
* Grade IV NYHA heart failure
* Prior clinical diagnosis of dementia
* Recent hospitalization for major illness or elective surgery (within 4 weeks)
* Terminal illness
* Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
* Subjects who are participating in ongoing RCTs of therapeutic interventions (including CTIMPs)
* Plan to move out of the region in which the trial is being conducted within the next 2 years (proposed minimum follow-up period)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 145 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in bone mineral density (BMD) | baseline and one year follow up

SECONDARY OUTCOMES:
Change in bone biomarkers | baseline and one year follow up
Bone mineral density (BMD) | 1 year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Rodondi, MD MAS, Principal Investigator — Clinic for General Internal Medicine, Bern University Hospital Bern
Locations (2):
- Switzerland (2):
  - Department of General Internal Medicine, Lausanne, Canton of Vaud
  - Clinic for General Internal Medicine, Bern University Hospital Bern, Bern

REFERENCES:
- [Background] Rodondi N, den Elzen WP, Bauer DC, Cappola AR, Razvi S, Walsh JP, Asvold BO, Iervasi G, Imaizumi M, Collet TH, Bremner A, Maisonneuve P, Sgarbi JA, Khaw KT, Vanderpump MP, Newman AB, Cornuz J, Franklyn JA, Westendorp RG, Vittinghoff E, Gussekloo J; Thyroid Studies Collaboration. Subclinical hypothyroidism and the risk of coronary heart disease and mortality. JAMA. 2010 Sep 22;304(12):1365-74. doi: 10.1001/jama.2010.1361. PMID 20858880
- [Background] Rodondi N, Newman AB, Vittinghoff E, de Rekeneire N, Satterfield S, Harris TB, Bauer DC. Subclinical hypothyroidism and the risk of heart failure, other cardiovascular events, and death. Arch Intern Med. 2005 Nov 28;165(21):2460-6. doi: 10.1001/archinte.165.21.2460. PMID 16314541
- [Derived] Buchi AE, Feller M, Netzer S, Blum MR, Gonzalez Rodriguez E, Collet TH, Del Giovane C, van Heemst D, Quinn T, Kearney PM, Westendorp RGJ, Gussekloo J, Mooijaart SP, Hans D, Bauer DC, Rodondi N, Aeberli D. Bone geometry in older adults with subclinical hypothyroidism upon levothyroxine therapy: A nested study within a randomized placebo controlled trial. Bone. 2022 Aug;161:116404. doi: 10.1016/j.bone.2022.116404. Epub 2022 Apr 2. PMID 35381390
- [Derived] Gonzalez Rodriguez E, Stuber M, Del Giovane C, Feller M, Collet TH, Lowe AL, Blum MR, van Vliet NA, van Heemst D, Kearney PM, Gussekloo J, Mooijaart S, Westendorp RGJ, Stott DJ, Aeberli D, Bauer DC, Hans D, Rodondi N. Skeletal Effects of Levothyroxine for Subclinical Hypothyroidism in Older Adults: A TRUST Randomized Trial Nested Study. J Clin Endocrinol Metab. 2020 Jan 1;105(1):dgz058. doi: 10.1210/clinem/dgz058. PMID 31702015